CLINICAL TRIAL: NCT06511375
Title: Comparative Effects of Sprint and Power Training on Speed and Repeated Sprint Ability in Cricket Fast Bowlers
Brief Title: Comparative Effects of Sprint and Power Training in Cricket Fast Bowlers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR &AHS/23/0476
Record Dates: First submitted 2024-06-11; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Sports Physical Therapy
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sprint training (Experimental): group 1 will perform sprint training for 4 weeks, 3 sessions per week
  Participants will perform 6 maximal 25-m sprint with recovery period of 25 seconds after each sprint for four weeks and three sessions per week.
  Participants will perform 10 m sprint 2 trials with 2 minutes recovery period between each trial for four weeks and three sessions per week.
  Participants will perform Vertical jump, 2 trials with 1-minute recovery period between each trial for four weeks, three sessions per week.
  Interventions: Other: sprint training
- power training (Experimental): GROUP 2 will perform POWER TRAINING for 4 weeks, 3 sessions per week Participants will perform Countermovement jump 2 trials, with 1-minute recovery between each trial for four weeks, three times per week.
  Participants will perform squat jump 2 trials with 1-minute recovery between each trial for four weeks, three times per week.
  Participants will perform broad jump 2 trials with 1-minute recovery between each trial for four weeks, three times per week.
  Interventions: Other: Power Training

INTERVENTIONS:
Other: sprint training — sprint training involves 20 meters sprint power training involve countermovement jump, squat jump and broad jump
  Arms: sprint training
Other: Power Training — GROUP 2 will perform POWER TRAINING for 4 weeks, 3 sessions per week Participants will perform Countermovement jump 2 trials, with 1-minute recovery between each trial for four weeks, three times per week.
  Participants will perform squat jump 2 trials with 1-minute recovery between each trial for four weeks, three times per week.
  Participants will perform broad jump 2 trials with 1-minute recovery between each trial for four weeks, three times per week.
  Arms: power training

SUMMARY:
Sprints can be a really effective way to improve participants cardiovascular fitness, strength and power, and running economy. Participants can gain bigger improvements and in less time with sprinting than with continuous easy running. Power training typically involves exercises which apply the maximum amount of force as fast as possible. Both these trainings are vital to increase the speed and repeated sprint ability in cricket fast bowlers.

DETAILED DESCRIPTION:
Fast bowling requires a highly specialized and unique training approach as the whole body is used in the delivery of the ball to achieve maximum velocity. For this purpose, the fast bowlers must perform the sprint training which is high intensity interval training as it boosts the speed and power, helps to run faster, build muscles and increase the cardiovascular health. Along with sprint training fast bowlers undergo power training which also helps to run faster, improve strength and speed and maintain fitness.

It will be a Randomized clinical trial with sample size of 34 calculated by G-power with 10- m sprint test, using non probability convenient sampling technique. The study will include physically fit and healthy fast bowlers of age 18-30 years. Participants will be divided into 2 equal experimental groups. One group will perform sprint training which include 10 meter run or repeated sprint ability and other will perform power training including squat jump or countermovement jump consisting of 12 sessions for 4 weeks (3 sessions each week). Data will be assessed by using SPSS version 25

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18- 30 years
2. Fast bowlers (male and female)
3. Physically fit and healthy athletes
4. Players must have fast bowling experience of at least 2 years. -

Exclusion Criteria:

1. Fast bowlers with musculoskeletal conditions ( back pain, foot and ankle injuries, fracture of lower limb and bone deformity, patellar tendinopathy, ligamentous and meniscal injury)
2. Vestibular and visual disorders
3. cardiac and respiratory issues -

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-08-25 (Estimated)

PRIMARY OUTCOMES:
Speed | 10 months
  speed is assessed by 10-m sprint test. participants will run for 10 meters on the sound of GO. the time taken for the completion of 10 meter track will be recorded by a handled stopwatch. Measurements will be taken before and after 10-m sprint test.
Repeated Sprint Ability | 10 months
  Repeated-sprint ability (RSA) is now well accepted as an important fitness component in team-sport performance. It is broadly described as the ability to perform repeated short (~3-4 s, 20-30 m) sprints with only brief (~10-30 s) recovery between bouts. measurements will be taken before and after the repeated sprint ability test.

CONTACTS AND LOCATIONS:
Overall Officials: Amna Shahid, T-DPT, Principal Investigator — Riphah International University
Locations (1):
- Zafarwal playzone, Zafarwal, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No